CLINICAL TRIAL: NCT05486871
Title: Oncological and Functional Outcomes of Laparoscopic Partial Nephrectomy in Renal Cell Carcinoma Stages T1 Versus T2a: Prospective Comparative Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Attia, assistent lecturer at urology department, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-07-20
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- renal cell carcinoma stages T1 (Active Comparator): laparoscopic partial nephrectomy in renal cell carcinoma stage T1
  Interventions: Procedure: laparoscopic partial nephrectomy
- renal cell carcinoma stages T2a (Active Comparator): laparoscopic partial nephrectomy in renal cell carcinoma stage T2a
  Interventions: Procedure: laparoscopic partial nephrectomy

INTERVENTIONS:
Procedure: laparoscopic partial nephrectomy — This is a prospective non- randomized controlled study of patients with RCC Who will be referred to urology department, Sohag university hospital. Our comparative study contained two groups according to tumor stage at preoperative contrast study:
  Group [A] : 15 patients with T1 RCC (≤ 7 cm). Group [B] : 15 patients with T2a RCC (≤ 10 cm). the patients will be subjected to laparoscopic partial nephrectomy then will be followed up for two years for oncological and functional outcomes.

SUMMARY:
RCC represents around 3% of all cancers, with the highest incidence occurring in Western countries . Within the several RCC risk factors identified, smoking, obesity, and hypertension are most strongly associated with RCC .

The EUA guidelines recommend PN for patients with T1 tumors, as PN preserved kidney function better after surgery, thereby potentially lowering the risk of development of cardiovascular disorders as well as improving overall survival(OS) for PN compared to RN, there is very limited evidence on the optimal surgical treatment for patients with larger renal masses (T2) .

Currently, the upper limit of PN indications remains undefined and is determined by an individual surgeon's expertise and preference. The degree of variability in the choice between PN and RN for a given tumor increases with tumor size. Surgeons committed to nephron-sparing are likely to expand the indications of PN, while those concerned with increased morbidity and doubtful of the clinical relevance of a moderate decrease in renal function are likely to perform RN, regardless of tumor size .

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized RCC ≤ 10 cm in preoperative contrast enhanced imaging(T1 and T2a).

Exclusion Criteria:

* Patients who had other tumors
* benign tumors
* clinically unfit
* metastatic RCC
* patients with Clinical T2b or higher tumors,
* tumors with maximum diameter > 10cm

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Renal function. | 3month
  Patients' pre and postoperative eGFR values were calculated using the Chronic Kidney Disease Epidemiology Collaboration equation, with the postoperative eGFR based on the creatinine measurement taken closest to 1 yr after surgery (between 9 and 15 month postoperatively). The eGFR downgrade was defined as preoperative eGFR 60 ml/min/1.73 m2 and postoperative eGFR <60 ml/min/1.73 m2 at 1 yr after surgery.
Post-operative complications. | 3 month
  complications within 90 days of operation were prospectively collected and classified based on the modified Clavien -Dindo grading system
Local recurrence. | 3 month
  radiological investigation in the form of contrast enhanced CT abdomen and pelvis or MRI incase of raised serum creatinine
Distant metastases. | 3 month
  radiological investigation in the form of contrast enhanced CT abdomen and pelvis or MRI incase of raised serum creatinine and bone scan incase of bone pain or pathological fractures CT BRAIN incase of manifestation of increased intracranial tension

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferlay J, Colombet M, Soerjomataram I, Dyba T, Randi G, Bettio M, Gavin A, Visser O, Bray F. Cancer incidence and mortality patterns in Europe: Estimates for 40 countries and 25 major cancers in 2018. Eur J Cancer. 2018 Nov;103:356-387. doi: 10.1016/j.ejca.2018.07.005. Epub 2018 Aug 9. PMID 30100160
- [Background] Vilaseca A, Guglielmetti G, Vertosick EA, Sjoberg DD, Grasso A, Benfante NE, Nguyen DP, Corradi RB, Coleman J, Russo P, Vickers AJ, Touijer KA. Value of Partial Nephrectomy for Renal Cortical Tumors of cT2 or Greater Stage: A Risk-benefit Analysis of Renal Function Preservation Versus Increased Postoperative Morbidity. Eur Urol Oncol. 2020 Jun;3(3):365-371. doi: 10.1016/j.euo.2019.04.003. Epub 2019 Apr 30. PMID 31411969
- [Background] Munoz-Rodriguez J, Prera A, Dominguez A, de Verdonces L, Rosado MA, Martos R, Prats J. Laparoscopic partial nephrectomy: Comparative study of the transperitoneal pathway and the retroperitoneal pathway. Actas Urol Esp (Engl Ed). 2018 May;42(4):273-279. doi: 10.1016/j.acuro.2017.09.008. Epub 2017 Nov 21. English, Spanish. PMID 29169703
- [Background] Capitanio U, Bensalah K, Bex A, Boorjian SA, Bray F, Coleman J, Gore JL, Sun M, Wood C, Russo P. Epidemiology of Renal Cell Carcinoma. Eur Urol. 2019 Jan;75(1):74-84. doi: 10.1016/j.eururo.2018.08.036. Epub 2018 Sep 19. PMID 30243799